CLINICAL TRIAL: NCT03036670
Title: Eosinophilic Granulomatosis With Polyangiitis Cohort
Acronym: EGPA Cohort
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2015/130
Record Dates: First submitted 2016-09-26; First posted 2017-01-30 (Estimated); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Churg-Strauss Syndrome
MeSH Terms: conditions — Churg-Strauss Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
EGPA (Eosinophilic Granulomatosis with Polyangiitis, previously Churg-Strauss syndrome) is a rare vasculitis, characterised by asthma, rhinosinusitis and eosinophilia. There has previously been confusion around diagnostic criteria, with multiple sets of classification criteria being used inappropriately for diagnosis. The ERS formed a taskforce to produce specific diagnostic criteria, and these divided the Churg-Strauss Syndrome cohort into two groups - vasculitic EGPA and tissular Hypereosinophilic Asthma with Systemic Manifestations (HASM). It is not known if the groups separated by the diagnostic criteria are also separated in clinical symptomatology, or if their disease course varies, and this could have significant impact on management and further research.

DETAILED DESCRIPTION:
Background Eosinophilic Granulomatosis with Polyangiitis (EGPA, previously Churg-Strauss Syndrome) is a rare, idiopathic, ANCA associated vasculitis (AAV), alongside Granulomatosis with Polyangiitis (GPA) and Microscopic Polyangiitis (MPA). It is an eosinophilic small/medium vessel vasculitis characterised by asthma, rhinosinusitis and eosinophilia. Patients can also suffer renal, cardiac, gastrointestinal and neurological involvement. First described by Churg and Strauss in 1951, exact epidemiology remains difficult because of a lack of clear diagnostic criteria. It appears to have a prevalence of around 11-13 per million population with a mean age of 50 years old and represents 10% of diagnosed vasculitides.

Following Churg and Strauss' original paper, the first attempt to provide diagnostic clarity was provided by John Lanham in 1984. Lanham listed symptoms seen in a set of patients with EGPA and suggested which symptoms were required for the disease and which symptoms were "additional". The American College of Rheumatology (ACR) in 1990 published a list of 6 symptoms to assist with classification of vasculitides, created by comparing 20 patients with EGPA with 787 patients with other forms of vasculitis. This was frequently used for diagnosis despite being intended for classification. In 1994, and revised in 2012, the International Chapel Hill Consensus Conference produced a nomenclature and definition for vasculitides, again frequently incorrectly used as diagnostic criteria. Finally, in 2014, diagnostic criteria were provided by the European Respiratory Society Churg Strauss Syndrome (ERS-CSS) taskforce; however published literature still uses a variety of criteria.

EGPA is recognised as a Th2 predominant disease with elevated levels of IL-4, IL-5, IL-13 and IgE according to a number of case control studies and case reports. Association between IL-10 levels and ANCA negative EGPA has been reported. Th17 responses also seem to be elevated with raised serum IL-25 reported, potentiating Th2 cytokine release. Eosinophil products are detectable in serum, BAL, urine and biopsies with varying time-courses. Roles of other cells such as regulatory T cells, memory T cells, dendritic cells, macrophages, ILCs and others are being investigated.

Previous work within the investigators' unit has demonstrated disturbances in the coagulation system in patients with asthma. The investigators have demonstrated that, while moderate asthma appears to favour fibrinolysis, severe asthma is a fibrinogenic condition. Deposition of fibrin within the airways in fatal asthma has been previously recognised, but a case study demonstrated strong activation of the coagulation system five days prior to an exacerbation. Another case study has demonstrated increased activation of the coagulation system in a patient with active EGPA which normalised on remission, but more in depth work has not been done.

It has been previously recognised that ANCA positive patients often have a different disease phenotype to those who are ANCA negative, suffering with more vasculitic symptoms and renal disease but less cardiac involvement. In 2014 the ERS-CSS taskforce provided diagnostic criteria for these two main phenotypes - separating the vasculitic phenotype which remains called Eosinophilic Granulomatosis with Polyangiitis (EGPA), from the ANCA negative tissular phenotype called Hypereosinophilic Asthma with Systemic Manifestations (HASM). It is currently unclear if this distinction matches biological endotypes, or whether different treatment strategies are advisable between the two groups. It is possible that HASM is a precursor state to full vasculitic EGPA, however the increased incidence of cardiac manifestations within this group would point away from this, as would the differing prevalence of genetic markers such as IL-10 promoter activation.

Prior to the advent of corticosteroid use, prognosis of EGPA was poor with a mortality rate of 50% at 3 months. Treatment primarily consists of immunosuppression with corticosteroids, with induction therapy using cyclophosphamide in severe cases. Rituximab is approved for use in GPA and MPA, while case reports demonstrate a good effect in patients with severe, refractory EGPA, uncontrolled on other therapy. Those who suffer from CSS can be exposed to prolonged steroid therapy with the majority of patients experiencing side effects of their medication such as weight gain, osteopaenia, impaired glucose tolerance, cataracts and skin atrophy. Steroid sparing agents such as azathioprine and mycophenolate are used with variable effect. Treatment is primarily guided by eosinophil count and symptom scores such as the Birmingham Vasculitis Activity Score (BVAS) as there are not currently any diagnostic tests or EGPA-specific biomarkers. Presence of a specific biomarker would allow more accurate alterations in patients' mediation, as non-specific symptoms can imitate EGPA and prompt increases in steroid doses.

Research questions Do the ERS-CSS diagnostic criteria divide the PHT cohort into groups with distinct clinical characteristics? How do the EGPA and HASM groups differ in clinical and physiological characteristics and how do these change over time?

Potential impact If the investigators confirm that EGPA and HASM represent distinct clinical entities within our cohort, further research into biological mechanisms and treatment options is needed, and this work will help to guide further studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or above.
* Cared for currently or previously cared for at Portsmouth Hospitals NHS Trust
* Diagnosed with EGPA/HASM according to clinicians

Exclusion Criteria:

- Medical notes not obtainable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants are adults with Churg-Strauss syndrome under the care of Portsmouth Hospitals NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis according to various diagnostic criteria | From date of diagnosis for 5 years
  The diagnosis of each participant according to different diagnostic or classification criteria (ERS-CSS, Chapel Hill, ACR, Lanham) based on all test results available between the point of diagnosis and 60 months later

SECONDARY OUTCOMES:
Corticosteroid dose | From date of diagnosis for 5 years
  Stable doses (taken for ≥4 weeks) of oral and inhaled corticosteroids at diagnosis and 12 monthly up to 5 years
Immunosuppressive medication | From date of diagnosis for 5 years
  Which additional immunosuppressive medication had been given and when
Comorbid conditions | From date of diagnosis for 5 years
  List of comorbidities
Biopsy findings | From date of diagnosis for 5 years
  List of Biopsy results
Relapse rates | From date of diagnosis for 5 years
  Rate of relapses or flares
Peak disease activity | From date of diagnosis for 5 years
  maximum disease activity from diagnosis to 5 years as defined by BVAS score and VDI score

CONTACTS AND LOCATIONS:
Overall Officials: Anoop J Chauhan, PhD FRCP, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom